CLINICAL TRIAL: NCT03981354
Title: Prognostic Potential of the Preoperative Nutritional Status and Its Postoperative Variation in Patients Undergoing Hip Arthroplasty
Brief Title: Nutritional Status and Its Modifications After Hip Replacement
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: NUTRIANCA (PI: M Briguglio); L4133 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2019-05-22; First posted 2019-06-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hip Arthropathy; Malnutrition; Anemia; Frail Elderly Syndrome
MeSH Terms: conditions — Malnutrition; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data literature lacks of evidence concerning the variation of the nutritional status in patients undergoing hip surgery, thus preventing an effective application a nutritional support program. It is therefore necessary to start identifying the clinical steps (pre-operative and post-operative) that may be defined as critical control points for malnutrition. The observation should foresee the identification of nutritional status indicators, such as weight, hemoglobin, albumin, food intake, and others that might affect a proper recovery. This study aims to investigate the prognostic nutritional factors that might influence clinical outcomes, and their variation in relation to hospitalization and rehabilitation periods.

DETAILED DESCRIPTION:
Data literature lacks of evidence concerning the variation of the nutritional status in patients undergoing hip surgery, thus preventing an effective application a nutritional support program. It is therefore necessary to start identifying the clinical steps (pre-operative and post-operative) that may be defined as critical control points for malnutrition. Patients undergoing hip surgery would be enrolled before the surgical operation and would be evaluated three times: preoperative, postoperative, and after discharge. The observation should foresee the identification of nutritional status indicators, such as weight, hemoglobin, albumin, food intake, and others that might affect a proper recovery. This study aims to investigate the prognostic nutritional factors that might influence clinical outcomes, and their variation in relation to hospitalization and rehabilitation periods.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* arthroplasty intervention program with hip prosthesis placement
* signature and acceptance of informed consent to collaborate in all the procedures necessary for the study

Exclusion Criteria:

* heart failure stage III-IV
* renal failure stage III-IV
* actual cancer
* past neurological disorders (including, but not limited to cerebral ischemia, cerebral haemorrhages, brain tumors, endocranial aneurysms)
* neurodegenerative disorders (including, but not limited to Alzheimer's dementia, fronto-temporal dementia)
* actual major psychopharmacological therapies
* pregnancy certified by self-declaration
* inability to adhere to the rehabilitation protocol or to carry out the controls
* non-acceptance of informed consent
* revision interventions
* previously established and documented sleep disorders
* shift or part-time worker

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of hemoglobin at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  One of the main decision-making factors that guide the clinician to discharge the patient is the hemoglobin level. The association between preoperative hemoglobin and hemoglobin at discharge was already observed in past orthopedic cohorts, with a loss of 3.3 g/dl being considered clinically relevant. Patients with a better nutritional status may have a reduced fall in hemoglobin after the surgical operation.

SECONDARY OUTCOMES:
Change from baseline level of pre-albumin at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Pre-albumin (mg/dl)
Change from baseline level of total lymphocyte count at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Total lymphocyte count (cells/mm^3)
Change from baseline level of iron at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Iron (μg/dl)
Change from baseline level of vitamin D at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  25[OH]D (ng/ml)
Change from baseline of weight 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Weight (kg)
Change from baseline of calf circumference 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Calf circumference (cm)
Change from baseline of % of fat mass at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Bioelectrical impedance analysis (% of fat mass and % of lean mass)
Change from baseline of hand-grip strength at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Hand-grip strength (kg). For this test, the higher values, the better is.
Change from baseline of FIM test at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Functional Independence Measure (FIM) (18-126 point scale). For this test, the higher values, the better is.
Change from baseline of 10 meter walking test at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  10 meter walking test (m/s). For this test, the higher values, the better is.
Change from baseline of POMA at 14 days after surgical operation | Before the surgical operation, after 3 days, after 14 days.
  Performance Oriented Mobility Assessment (POMA) (0-32 point scale). For this test, the higher values, the better is.

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided